CLINICAL TRIAL: NCT04806295
Title: The Leukemia and Lymphoma Society (LLS) National Research Registry
Status: Recruiting | Type: Observational
Sponsor: Blood Cancer United (Other)
Responsible Party: Sponsor
Other Study IDs: LLSNRR-17-001
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Blood Cancer
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: any/all treatments for blood cancer — Following people undergoing any/all treatments for blood cancer.

SUMMARY:
The Leukemia and Lymphoma Society (LLS) has built a National Research Registry to evaluate real world experiences and medical outcomes for people with blood cancer, before, during, and after blood cancer treatments.

DETAILED DESCRIPTION:
The LLS National Research Registry is a real-world experiences and outcomes research registry; a collection of patient information and medical data, over time, about people who have a particular disease or condition, or who receive a particular treatment.

The LLS National Research Registry Protocol will:

1. Answer research questions using data collected from people with blood cancers. Such research involves analyses of subject profile information completed by subjects and medical records data.
2. Obtain permission from LLS National Research Registry research subjects to have Ciitizen, a third-party engaged by LLS, act as their proxy to retrieve full medical record data including images at no cost to research subjects. Note: Patient can choose to upload their medical records into their account, directly.
3. Obtain permission from LLS National Research Registry research subjects to share summary data with research partners (like academic researchers, advocacy groups, and pharmaceutical companies) that are advancing treatments for blood cancer. "Summary data" represents the important elements of medical record data, coded for research use, with personal identifiers like name, address, and phone number removed.
4. Obtain permission from LLS National Research Registry research subjects to be contacted from time to time, for them to provide updated medical information.

ELIGIBILITY:
Inclusion Criteria:

People with blood cancer, before, during, and after blood cancer treatments.

Exclusion Criteria:

People unable or unwilling to sign informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with blood cancer, before, during, and after blood cancer treatments.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-07-24 (Actual); Primary Completion 2027-07-23 (Estimated); Study Completion 2027-07-23 (Estimated)

PRIMARY OUTCOMES:
LLS will monitor outcomes of people being treated for blood cancer. | 10 years
  . The LLS National Research Registry will collect data on up to 1000 research subjects, over up to 10 years, storing that data, including protected health information (PHI) and images, in secure databases, and share de-identified summary data with research partners (like academic researchers, advocacy groups, and pharmaceutical companies) that are advancing treatments for blood cancer. Participation in The LLS National Research Registry may not give research subjects any immediate benefit. It is hoped the knowledge gained from data collected in The LLS National Research Registry will benefit people with blood cancers in the future using this information for research purposes, directed at blood cancers and associated comorbidities.

CONTACTS AND LOCATIONS:
Locations (1):
- Lymphoma and Leukemia Society, Rye Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Participating subjects will be asked to provide permission to share de-identified summary data with research partners (like academic researchers, advocacy groups, and pharmaceutical companies) that are advancing treatments for cancer, neurological disorders, and other diseases. "Summary data" represents the important elements of medical record data, coded for research use, with personal identifiers like name, address, and phone number removed.
Supporting Information: Study Protocol
Time Frame: As data is collected, de-identified and stored in a secure database, it will be provided over time to LLS investigators and investigators approved by LLS.
Access Criteria: De-identified data will be made available to LLS investigators and investigators approved by LLS.